CLINICAL TRIAL: NCT03343665
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of Nivolumab at the Fixed Dose 40 mg (Nivo40) in Patients With Relapsed or Refractory Hodgkins Lymphoma.
Brief Title: Treatment With Nivolumab at the Fixed Dose 40 mg (Nivo40) in Patients With Relapsed/Refractory Hodgkins Lymphoma
Acronym: Nivo40
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: №30/17-н
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hodgkin Lymphoma
Keywords: Nivolumab
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab 40 mg (Experimental): Experimental: Nivolumab Nivolumab 40 mg IV over 60 minutes on day 1. Treatment repeats every 14 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab 40 mg in 4 ml Injection

INTERVENTIONS:
Drug: Nivolumab 40 mg in 4 ml Injection — 40 mg by intravenous (IV) infusion on day 1 Duration of cycle 14 days
  Other Names: Opdivo

SUMMARY:
A phase I/II trial to evaluate the safety and efficacy of nivolumab at the fixed dose 40 mg in patients with relapsed or refractory Hodgkins lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed Hodgkins lymphoma
* Relapsed or refractory disease after at least two prior lines of treatment
* Age 18-70 years old
* Signed informed consent
* No severe concurrent illness

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 months
  Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by LYRIC criteria

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).
Duration of Response (DOR) | 12 months
Progression-Free Survival (PFS) | 12 months
Overall Survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris V Afanasyev, Ph.D, Principal Investigator — St. Petersburg State Pavlov Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lepik KV, Fedorova LV, Kondakova EV, Zalyalov YR, Babenko EV, Lepik EE, Kotselyabina PV, Beynarovich AV, Popova MO, Volkov NP, Stelmakh LV, Baykov VV, Moiseev IS, Mikhailova NB, Kulagin AD, Afanasyev BV. A Phase 2 Study of Nivolumab Using a Fixed Dose of 40 mg (Nivo40) in Patients With Relapsed/Refractory Hodgkin Lymphoma. Hemasphere. 2020 Sep 23;4(5):e480. doi: 10.1097/HS9.0000000000000480. eCollection 2020 Oct. PMID 33062947